CLINICAL TRIAL: NCT04272606
Title: Prospective, Randomized, Double Blind Study on the Effects of Tranexamic Acid on Intraoperative Blood Loss During Lumbar Spinal Fusion And Instrumentation
Brief Title: TXA in Spinal Fusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catherine R. Olinger (Other)
Responsible Party: Sponsor-Investigator, Catherine R. Olinger, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201912099
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Degenerative Disc Disease
Keywords: Posterior Lumbar Interbody Fusion; Transforaminal Lumbar Interbody Fusion; Tranexamic Acid; Neurosurgery; Delirium
MeSH Terms: conditions — Intervertebral Disc Degeneration; Delirium | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Phase 2B randomized, single-center, double-blinded, placebo vs treatment clinical trial with 1:1 randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): 1:1 randomization, given tranexamic acid during surgery, visual acuity exam
  Interventions: Drug: Tranexamic Acid; Diagnostic Test: Visual Acuity Exam; Diagnostic Test: 3 Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM)
- Placebo (Placebo Comparator): 1:1 randomization, given standard of care treatment during surgery, visual acuity exam
  Interventions: Drug: Saline Solution; Diagnostic Test: Visual Acuity Exam; Diagnostic Test: 3 Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM)

INTERVENTIONS:
Drug: Tranexamic Acid — Antifibrinolytic Agent
  Other Names: Cyklokapron
  Arms: Treatment
Drug: Saline Solution — Placebo
  Arms: Placebo
Diagnostic Test: Visual Acuity Exam — Supplemented into standard of care daily neurological exam on day of surgery and day after
  Other Names: Eye Exam
Diagnostic Test: 3 Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) — 3D-CAM is a brief verbal assessment tool that can be used to test patients and study patients for delirium.

SUMMARY:
Tranexamic acid and placebo will be given during surgery to patients who have elected to undergo lumber interbody fusion on 2 or more levels. Information regarding blood loss, transfusions needed, postoperative cognitive status (including delirium), postoperative markers of systemic inflammation and duration of hospital stay will be collected.

DETAILED DESCRIPTION:
This study is to assess whether tranexamic acid (a drug that is used to coagulate the blood and reduce bleeding) use in lumbar spinal fusion can reduce blood loss and postoperative delirium compared to placebo. Thusly reducing need for transfusion, shorting the hospital stay and improving outcomes. For this the study will randomize patients who are receiving elective lumbar interbody fusion (PLIF or TLIF) of 2 or more levels for degenerative disc disease (DDD) into 2 groups. Group 1 would receive tranexamic acid during the surgery while group 2 will receive placebo. Blood loss during the surgery and postoperatively (while the patient has a drain) will be monitored along with the amount of transfusions needed, postoperative cognitive status (including delirium), postoperative markers of systemic inflammation, and and the duration of hospital stay. Delirium occurrence and severity will be assessed daily for the first 5 days after surgery or at discharge, whichever comes first. Cognitive status (neuropsychological tests) will be assessed at post-discharge follow up visits and compared to preoperative status.

The drug or placebo are only given during the surgery. The patient population includes elective cases of patient undergoing lumbar spinal fusion of 2 or more levels. Spinal fusions are known to be associated with blood loss, especially when the surgeries are long and more levels need to be fused.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-90 years
2. American Spinal Injury Association (ASA) Impairment Scale anesthesia risk of I to IV
3. Patients undergoing 2 or more levels of posterior lumbar interbody fusion for DDD. This includes PLIF or TLIF.
4. Patients have failed conservative management, which include physical therapy (PT) or occupational therapy (OT) and/or injections.

Exclusion Criteria:

1. ASA class V
2. Patient unable to consent
3. Patient with chronic kidney disease stage III or above: baseline plasma creatinine>1.5mg/dL
4. Patient with known liver failure
5. Patients on anticoagulation or dual antiplatelets (presence of vascular stents).
6. Patients with artificial valves.
7. Patients with allergy to TXA
8. Patients with platelet count < 150 000,
9. Patients with PT>15s
10. Patients with Activated Partial Thromboplastin Time (APPT) >38s
11. History of stroke or (an) unprovoked thromboembolic event(s).
12. History of intracranial bleeding,
13. Pregnancy
14. known defective color vision
15. history of venous or arterial thromboembolism or active thromboembolic disease
16. Patients with severe pulmonary or cardiac disease.
17. Patients who refuse transfusion of blood products
18. Patients with chronic anemia with Hg<8
19. Patients undergoing lumbar fusion for disease other than DDD (neoplasm)
20. Patients undergoing lumbar fusion by anterior or lateral approach.
21. Minimally invasive TLIF are excluded.
22. Emergent cases.
23. Women on hormonal contraception
24. Retinal vein or artery occlusion
25. Hypercoagulability
26. Seizure disorder
27. Current use of tretinoin
28. Current use of chlorpromazine
29. Breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Olinger, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hindman BJ, Olinger CR, Woodroffe RW, Zanaty M, Deifelt Streese C, Zacharias ZR, Houtman JCD, Wendt LH, Ten Eyck PP, O'Connell-Moore DJ, Ray EJ, Lee SJ, Waldschmidt DF, Havertape LG, Nguyen LB, Chen PF, Banks MI, Sanders RD, Howard MA 3rd. Exploratory randomised trial of tranexamic acid to decrease postoperative delirium in adults undergoing lumbar fusion-a trial stopped early. BJA Open. 2025 Apr 14;14:100403. doi: 10.1016/j.bjao.2025.100403. eCollection 2025 Jun. PMID 40276619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 123 subjects were enrolled and consented. Prior to randomization, 37 subjects were excluded and did not get randomized.
Pre-assignment Details: 37 subjects were excluded and not randomized due to the following reasons:
  * Exclusion criteria was found (14 subjects)
  * Surgery cancelled (8 subjects)
  * Subjects withdrew (5 subjects)
  * Surgery changed to min invasive and so subject did not qualify (3 subjects)
  * Surgeon decision (2 subjects)
  * trial on hold during randomization period (2 subjects)
  * study medication order problems (3 subjects)
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 44 | 42
Completed | 43 | 40
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 21 | 47
  >=65 years | 17 | 19 | 36
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [52 to 72] | 63 [55 to 71] | 61 [54 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 23 | 18 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 43 | 37 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 40 | 38 | 78
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 40 | 83

OUTCOME MEASURES:

1. Primary Outcome: Transfusion
Description: The number of participants who had red blood cells (RBC) transfused:
  1. Intraoperatively
  2. Postoperatively (prior to discharge or at day 5, whichever occurred first)
  3. Either Intraoperatively or Postoperatively
Time Frame: Assessed up to 5 days or until discharge, whichever came first, data collected on discharge day or day 5 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 43 | 40
Participants
  Intraoperatively | 7 | 6
  Postoperatively (prior to discharge or at day 5, whichever occurred first) | 9 | 8
  Either Intraoperatively or Postoperatively | 10 | 10

2. Primary Outcome: Blood Loss
Description: Amount of blood loss:
  1. Intraoperatively
  2. Postoperatively (prior to discharge or at day 5, whichever occurred first)
  3. Either Intraoperatively or Postoperatively
Time Frame: Assessed up to 5 days or until discharge, whichever came first, data collected on discharge day or day 5 reported
Measure: Median (Inter-Quartile Range); unit: ml per instrumented vertebral level
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 43 | 40
ml per instrumented vertebral level
  Intraoperatively | 167 [87 to 250] | 110 [67 to 176]
  Postoperatively (prior to discharge or at day 5, whichever occurred first) | 128 [97 to 186] | 207 [132 to 258]
  Either Intraoperatively or Postoperatively | 305 [186 to 412] | 333 [241 to 428]

3. Primary Outcome: Delirium Occurrence
Description: Delirium occurrence (yes/no) using daily 3D-CAM delirium assessment instrument.
Time Frame: Assessed up to 5 days or until discharge, whichever came first, data collected on discharge day or day 5 reported
Measure: Number; unit: participants with delirium
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 32 | 33
participants with delirium | 7 | 11

4. Secondary Outcome: Delirium Severity
Description: Severity (score 0-20) using daily 3D-CAM delirium assessment instrument. Minimum=0 (no delirium) Maximum=20 (worse delirium)
Time Frame: Assessed up to 5 days or until discharge, whichever came first, data collected on discharge day or day 5 reported
Measure: Median (Inter-Quartile Range); unit: 3D-CAM Points
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 32 | 33
3D-CAM Points | 1.10 [0.48 to 2.50] | 1.00 [0.50 to 2.00]

5. Secondary Outcome: Change in Interleukin-6 Concentration.
Description: Measure of systemic inflammation using Interleukin-6 change between preoperative and 24 postoperatively blood draw.
Time Frame: Preoperatively and 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: pg per ml
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 16 | 15
pg per ml | 25.7 [11.3 to 35.8] | 10.6 [5.3 to 68.2]

6. Secondary Outcome: Length of Postoperative Stay Prior to Discharge
Description: Length of postoperative stay prior to discharge in days
Time Frame: Days thru day of discharge
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 43 | 40
Days | 3 [2 to 6] | 3 [2 to 5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on all subjects until their final postoperative follow up clinic visit (typically at or around 3 months).
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/43 | 2/40
Other Adverse Events (participants affected / at risk) | 6/43 | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=43) | Placebo (N=40)
Pulmonary Embolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Pulmonary embolism 22 days after surgery, after discharge. Determined not to be attributed to study participation.
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) — Embolic stroke 69 days after surgery, following discharge. Determined not to be attributed to study participation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=43) | Placebo (N=40)
Vision Change (Eye disorders) | 2 (2) | 0 (0) — Temporary, unexplained vision change. Not attributed to study participation.
Renal Dysfunction (Renal and urinary disorders) | 2 (2) | 4 (4) — Creatinine increase > 20% of baseline on post-operative day 1. All resolved and not attributed to study participation.
Wound Complication (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — Delayed wound healing. Not attributed to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT04272606/Prot_002.pdf
  • Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT04272606/SAP_003.pdf